CLINICAL TRIAL: NCT02396875
Title: Selective Coronary Vein Sampling in Dyssynchronous Heart Failure and Cardiac Resynchronisation Therapy to Assess Physiological Response to Exercise and Characterise Regional Release of Novel Biomarkers
Brief Title: Selective Coronary Vein Sampling in Left Bundle Branch Block and CRT
Acronym: MicroCRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14/LO/1765
Record Dates: First submitted 2014-10-24; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1 (Experimental): 40 patients undergoing CRT will have venous samples taken from two CS tributaries, peripheral venous and peripheral arterial sites at the time of CRT insertion at the time of device implant. Blood samples will be analysed for metabolites and novel biomarkers They will then undergo repeat sampling at 6 months to assess for changes in the biomarker profile including CS sampling.
  Interventions: Procedure: Central blood sampling pre and post CRT implant
- Group 2 (Active Comparator): A control arm of 15 patients with heart failure and no dyssynchrony will undergo peripheral venous sampling for novel biomarkers and this will be repeated at 6 months. These samples will allow for control against the dyssynchronous heart failure group and also for temporal changes in biomarker expression.
  Interventions: Procedure: Peripheral blood sampling
- Group 3 (Active Comparator): A control arm of 15 patients with normal hearts will undergo peripheral venous sampling for novel biomarkers and this will be repeated at 6 months. These samples will allow for control against the dyssynchronous heart failure group and also for temporal changes in biomarker expression.
  Interventions: Procedure: Peripheral blood sampling
- Group A (Experimental): 10 patients from Group 1
  On the day preceding the CRT implant will attend hospital for a temporary invasive catheter study. The patient will have a radial sheath positioned in the arterial system. A pacing protocol will be performed using a pacing wire inserted into the right atrium. Coronary sinus venous blood sampling will be performed using a catheter placed via the femoral or internal jugular vein. At the chief investigator's discretion a specially designed exercise bicycle that allow supine exercise in the catheter lab will be used rather than the atrial pacing wire.
  6 months post implant the patients will return to the catheter laboratory for a further study. This will repeat the protocol but with the device having been on for 6 months. This will require further study as described above.
  Interventions: Procedure: Blood sampling and exercise protocol pre and post CRT implant
- Group B (Active Comparator): 5 patients form Group 2.
  Patients will undergo a pacing or exercise protocol and have venous, coronary sinus and arterial blood sampled. They will revert to Group 2 for 6 month follow up
  Interventions: Procedure: Central blood sampling on one occasion and exercise protocol and 6 month peripheral sampling
- Group C (Active Comparator): 5 patients form Group 3
  Patients will undergo a pacing or exercise protocol and have venous, coronary sinus and arterial blood sampled. They will revert to Group 3 for 6 month follow up
  Interventions: Procedure: Central blood sampling on one occasion and exercise protocol and 6 month peripheral sampling

INTERVENTIONS:
Procedure: Blood sampling and exercise protocol pre and post CRT implant
  Arms: Group A
Procedure: Peripheral blood sampling
  Arms: Group 2; Group 3
Procedure: Central blood sampling pre and post CRT implant
  Arms: Group 1
Procedure: Central blood sampling on one occasion and exercise protocol and 6 month peripheral sampling
  Arms: Group B; Group C

SUMMARY:
Cardiac resynchronisation therapy (CRT) prolongs the life and improves the symptoms in patients with heart failure and electrical dyssynchrony. 30-50% of patients do not improve with the treatment which is both expensive and not without complication. Despite much research, we cannot accurately predict who will not respond. Furthermore, most heart failure patients gets symptoms on exercise and most studies have examined patients at rest. We propose to investigate the effect of exercise on different parts of the left ventricle by sampling various biomarkers of metabolism, myocardial injury and gene expression. We will then repeat the protocol following device insertion to look for changes. This novel work will require a small cohort of patients with heart failure and no electrical dyssynchrony and normal patients to act as controls. We will also measure novel biomarkers at different venous sites relating to different parts of the myocardium to determine whether they can be used to prognosticate or even predict response to CRT.

DETAILED DESCRIPTION:
We propose to examine the acute effects of exercise on patients with dyssynchronous electrical activation of the heart and heart failure and to compare the release of novel biomarkers in selective areas of coronary venous drainage by direct cannulation of different veins via the coronary sinus (CS).

The study design will separate patients into a minimally invasive arm (MINARM)and an invasive arm (INARM). The INARM will be recruited from patients in the MINARM.

MINARM

Group 1: 40 patients scheduled for CRT implant Group 2: 15 patients with heart failure and no dyssynchrony Group 3: 15 patients with normal hearts

Group 1:

40 patient undergoing CRT will have venous samples taken from the CS, two CS tributaries, peripheral venous and peripheral arterial sites at the time of CRT insertion at the time of device implant. Blood samples will be analysed for metabolites and novel biomarkers

They will then undergo repeat sampling at 6 months to assess for changes in the micro RNA and biomarker profile including CS sampling.

Group 2 and 3

A control arm of 15 patients with heart failure and no dyssynchrony (Group 2) and 15 patients with normal hearts (Group 3) will undergo peripheral venous sampling for biomarkers and this will be repeated at 6 months. These samples will allow for control against the dyssynchronous heart failure group and also for temporal changes in micro RNA expression.

10 patient from Group 1 and 5 from Group 2 and 3 will be invited to from part of the INARM at the time of recruitment.

INARM study

Methods:

GROUP A 10 pts with heart failure and dyssynchronous ventricular contraction GROUP B 5 pts with heart failure and no electrical dyssynchrony schedule for either coronary angiography or electrophysiology study.

GROUP C 5 pts schedule for diagnostic coronary angiography or electrophysiology study with normal cardiac function

The exact details of the protocol will vary depending upon the Group:

GROUP A

1 On the day preceding the CRT implant will attend hospital for a temporary invasive catheter study. A pacing protocol will be performed using a pacing wire inserted into the right atrium. Coronary sinus venous blood sampling will be performed using a catheter placed via the femoral or internal jugular vein. At the chief investigator's discretion a specially designed exercise bicycle that allow supine exercise in the catheter lab will be used rather than the atrial pacing wire.

3 6 months post implant the patients will return to the catheter laboratory for a further study. This will repeat the protocol but with the device having been on for 6 months. This will require further arterial access as described above. This study should take approximately an hour.

GROUP B and C

It is common practice for these patients to have a coronary angiogram to exclude ischaemic heart disease as the cause of their heart failure or chest pain or to have electrophysiology study to determine the mechanism of arrhythmia. If their angiogram is normal,we will perform a pacing protocol (this will be required if they are attending for an electrophysiology study). This will require 2 femoral venous access sites (similar to standard electrophysiological study) to allow temporary atrial pacing and acquisition of blood samples from the coronary sinus. Following the invasive part of the study patients in Group B and C will fall back into Group 2 and 3 of MINARM and attend at 6 month for peripheral blood sampling.

ELIGIBILITY:
Inclusion Criteria:

Group 1/A:

-Scheduled for CRT implant

Group 2/B -Heart failure without electrical dyssynchrony.

Group B:

-Scheduled for angiography for clinical grounds

Group 3/C -Patients without known heart disease

Group C:

-Scheduled for clinical angiography and found to have normal coronary arteries

Exclusion Criteria:

* Pregnancy
* Moderate to severe aortic valve disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Levels of Various biomarkers measured from different coronary veins at rest and following exertion both pre CRT implant and at 6 months | 2 years
  Biomarkers and metabolites to be assessed include but are not limited to O2, lactate, glucose, CKMB, hs trop, galectin3, Soluble St2, Nt proBNP, cardiac myosin binding protein C, 10 different micro RNA associated with myocardial stress/damage

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas Hospital Trust, London, United Kingdom